CLINICAL TRIAL: NCT01856231
Title: Lifestyle Physical Activity for People With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Janet L. Larson, Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00038130
Record Dates: First submitted 2013-05-09; First posted 2013-05-17 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: COPD
Keywords: COPD; Physical activity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Intervention Model Description: Lifestyle physical activity self-efficacy
Oversight: Data Monitoring Committee: No

ARMS (1):
- 8 week group (Experimental): Lifestyle physical activity self-efficacy
  Interventions: Behavioral: Lifestyle physical activity - self-efficacy

INTERVENTIONS:
Behavioral: Lifestyle physical activity - self-efficacy — Subjects will come into an exercise lab 2 days per week and perform 10-20 minutes of walking, 13 strength training exercises, stretching and a behavioral intervention including goal setting, etc.

SUMMARY:
The purpose of this preliminary study is to examine the effects of a program that includes two-months of structured lab-based training. The proposed study will examine the effects of a lifestyle physical activity intervention designed to increase PA in people with moderate and severe COPD. The intervention includes a combination of (a) structured laboratory-based exercises with a behavioral intervention, (b) structured home-based exercises and (c) lifestyle physical activities performed at home. The subjects will be followed for a total of 18 weeks.

DETAILED DESCRIPTION:
People with chronic obstructive pulmonary disease (COPD) experience a gradual decline in physical activity (PA). Exercise training in a structured pulmonary rehabilitation program can generate substantial gains in functional capacity, but increases in functional capacity do not necessarily lead to improvements in daily PA. The proposed study will examine the effects of a lifestyle physical activity intervention designed to increase PA in people with moderate and severe COPD. The intervention includes a combination of (a) structured laboratory-based exercises with a self-efficacy enhancing intervention, (b) structured home-based exercises and (c) lifestyle physical activities performed at home. The intervention gradually transitions subjects from the structured laboratory-based exercises that focus on walking and circuit training to fully integrated lifestyle physical activities that integrate structured home-based exercises and lifestyle physical activities into daily life. The purpose of this preliminary study is to examine the effects of a program that includes two-months of structured lab-based training and subjects will be followed for a total of 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 55 years or older
* Moderate to severe COPD (FEV1 < 80% and > 30% predicted; FEV1/FVC <70%) as the primary health problem
* Sedentary (less than 30 minutes of moderate activity 3 days/week)

Exclusion Criteria:

* No acute exacerbations or major illnesses requiring hospitalization in the last 8 weeks.
* No history of other major lung diseases as primary pulmonary problem, history of a recent heart attack or recent onset of chest pains with activity or increasing episodes of chest pain (unstable angina).
* No other health problems or mobility problems that limit physical activity.
* No child bearing potential

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-08; Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Change in physical activity measured by accelerometry | During initial visit (week 1), at 6 or 10 weeks (depending on group placement), and at week 18
  Subjects wear two activity monitors for seven consecutive days (Actipal and Actigraph). The study will compare the subject's activity level at the three time points listed.

SECONDARY OUTCOMES:
Change in 6 minute walk test | During initial visit (week 1), at 6 or 10 weeks (depending on group placement), and at week 18
  Subjects complete a 6 minute walk test measuring the total distance he/she can walk in 6 minutes at the three time points listed.
Change in lower extremity function (Short Physical Performance Battery) | During initial visit (week 1), at 6 or 10 weeks (depending on group placement), and at week 18
  Subjects complete a performance test measuring balance, gait speed, and leg strength (using a chair stand test) at the three time points listed.
Change in dyspnea and fatigue (Pulmonary Functional Status and Dyspnea Questionnaire-Modified) | During initial visit (week 1), at 6 or 10 weeks (depending on group placement), and at week 18
  Subjects complete a questionnaire answering questions about their level of dyspnea in various daily activities at the three time points listed.
Change in physical activity measured by CHAMPS questionnaire | During initial visit (week 1), at 6 or 10 weeks (depending on group placement), and at week 18
  Subjects fill out a questionnaire of their perceived physical activity at the three time points listed.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Larson, PhD, Principal Investigator — University of Michigan - School of Nursing
Locations (1):
- University of Michigan - School of Nursing, Ann Arbor, Michigan, United States